CLINICAL TRIAL: NCT05537701
Title: Tissue Eosinophils in Non-Small Cell Lung Cancer (the TEN Study)
Acronym: TEN
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Anne Sibille, Principal investigator, Centre Hospitalier Universitaire de Liege
Other Study IDs: 2022/158
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to describe eosinophil infiltration in resected (early stage) NSCLC.

Secondary objectives are:

* to investigate the correlation of T-Eos and B-Eos in the aforementioned patient population;
* to investigate the correlation between T-Eos and overall & disease-free survival;
* to investigate the localization of T-Eos (periphery vs. center of the tumor lesions).

ELIGIBILITY:
Inclusion Criteria:

* Resected, early stage NSCLC between 01-01-2015 and 30-04-2022 with available tumour tissue

Exclusion Criteria:

* Inclusion in a clinical study contraindicating enrollment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resected, early stage NSCLC between 01-01-2015 and 30-04-2022 with available tumour tissue for analysis will be included.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of tumor associated tissue eosinophilia by immunohistochemistry and computerised quantification | October 2022

SECONDARY OUTCOMES:
to investigate the correlation of tissue (T)-Eos and blood (B)-Eos in the aforementioned patient population | December 2022
  Tissue and blood eosinophil correlation
to investigate the correlation between T-Eos and overall & disease-free survival | December 2022
  overall and disease-free survival
to investigate the localization of T-Eos (periphery vs. center of the tumor lesions) | December 2022
  tissue eosinophil localisation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No